CLINICAL TRIAL: NCT00541944
Title: Establishment of an Algorithm for a Clinical Classfication of Hypoosmolar Hyponatremia
Acronym: CONA
Status: Completed | Type: Observational
Sponsor: University of Wuerzburg (Other)
Responsible Party: Principal Investigator, Martin Fassnacht, I am only the successor of the PI of the study, Bruno Allolio, who unfortunately died in the meantime, University of Wuerzburg
Other Study IDs: Wue-CONA-33/07
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Hyponatremia
Keywords: hyponatremia; diagnosis and treatment of hyponatremia; classification of hyponatremia
MeSH Terms: conditions — Hyponatremia; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma and urine
Oversight: Data Monitoring Committee: No

SUMMARY:
The prospective clinical diagnosis of hyponatremia is often very difficult- but requirement for an appropriate and riskless treatment of hyponatremia. This study try to establish an algorithm handling a prospective clinical categorization of hyponatremia and approving together the start of an appropriate symptomatic therapy.

ELIGIBILITY:
Inclusion Criteria:

* hypoosmolar hyponatremia with serum sodium concentration ≤129 mmol/l and serum osmolality ≤ 280 mosm/kg;
* age > 18 years;
* letter of agreement.

Exclusion Criteria:

* gravidity and lactation;
* restricted decision-making-ability

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients treated in an University Hospital in Germany
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2007-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Establishment of an clinical algorithm to differentiate the different causes of hyponatremia | One year

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Allolio, MD, Principal Investigator — Universtiy of Wuerzburg
Locations (1):
- University of Wuerzburg, Würzburg, Germany

REFERENCES:
- [Derived] Fenske W, Stork S, Koschker AC, Blechschmidt A, Lorenz D, Wortmann S, Allolio B. Value of fractional uric acid excretion in differential diagnosis of hyponatremic patients on diuretics. J Clin Endocrinol Metab. 2008 Aug;93(8):2991-7. doi: 10.1210/jc.2008-0330. Epub 2008 May 13. PMID 18477658